CLINICAL TRIAL: NCT03856541
Title: A Phase I, Open Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SHR-A1403 With Intravenous Infusion in Patients With Advanced Solid Tumors
Brief Title: A Study of SHR-A1403 in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1403-I-101
Record Dates: First submitted 2019-02-13; First posted 2019-02-27 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2019-01

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumor; C-Met antibody drug conjugate; Safety; Pharmacokinetics
MeSH Terms: interventions — SHR-A1403

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1403 Dose Escalation (Experimental): SHR-A1403 given intravenously (IV).
  Interventions: Drug: SHR-A1403

INTERVENTIONS:
Drug: SHR-A1403 — SHR-A1403 is a humanized anti C-Met immunoglobulin G2 (IgG2) monoclonal antibody conjugated with microtubule inhibitor. SHR-A1403 is provided as the lyophilized powder,40 mg/vial.SHR-A1403 was given intravenously per 3 weeks at the day 1.Intravenous infusion over 30 min
  Other Names: HTI-1066

SUMMARY:
SHR-A1403 is a humanized IgG2, anti-C-Met monoclonal antibody conjugated to microtubule inhibitor (c-Met ADC).The aim of this study is to assess the safety and tolerability of SHR-A1403，to define the dose limited toxicity（DLT）and the maximum tolerated dose (MTD)，to evaluate the pharmacokinetics of SHR-A1403，to assess the antitumor activity of SHR-A1403 in patients with advanced solid tumors preliminarily and to recommend the reasonable dosage regimen of SHR-A1403 for the follow-up clinical trial.

DETAILED DESCRIPTION:
This study is a phase I clinical trial of single arm，open-label，dose escalation with single and multiple doses.The safety,PK and preliminary efficacy of SHR-A1403 were evaluated respectively in the patients with advanced solid tumors that have invalid standard treatment or no standard and effective treatment.SHR-A1403 is administered with intravenous infusion every three weeks (q3w) for a treatment cycle.Dose limiting toxicities (DLT) observation will end after 3 weeks from the start of study treatment(21 days). The dose escalation is designed by Modified Toxicity Probability Interval-2 Designs（mTPI-2) and will continue until an MTD or preliminary RP2D is identified. 3 patients are enrolled and observed in the initial dose. After completing the DLT assessment, the next decision of dose escalation will be performed according to the mTPI-2 detailed dose climbing/descending plan. After each decision, 3 other patients will be enrolled in the next phase of dose escalation until the maximum number of subjects specified in the study protocol or the dose escalation terminated by the Safety Monitoring Committee(SMC).

The study consists of 3 periods: Screening Period (up to 14 days before the first dose), Treatment Period, and Follow-up Period (up to 3 months after the last dose of study treatment).

The safety and tolerability of SHR-A1403 will be assessed by ongoing reviews of clinical laboratory tests, Eastern Cooperative Oncology Group (ECOG) performance status, physical examinations, vital signs, ECG, and adverse events (AEs) as defined by the current version of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE 4.03). Safety will be monitored throughout the study.

Response assessment will be performed by the end of Cycle 2 (6 weeks after the first infusion). Subsequently, post-dose tumor response evaluations will be performed every 6 weeks for the first 6 months, then by every 12 weeks thereafter, and at short-term follow up. For subjects who discontinue study treatment, tumor imaging should also be performed at end of therapy. Tumor imaging will be performed for all subjects as feasible (e.g., may not be able to be performed in subjects who withdraw consent or would not be performed in subjects who are lost to follow-up) until documented progression of disease, intolerable toxicity, initiation of a new antitumor therapy, withdrawal of consent, or the occurrence of death or end of study, whichever occurs first.

Blood samples collected pre-dose and post-dose will be analyzed for PK variables. In general, PK data analysis will include, but will not be limited to, time to maximal serum concentration (tmax), maximal serum concentration (Cmax), area under the curve from time 0 to Day 21 of Cycle 1 (AUC0-21d), and observed terminal half life (t1/2) in Cycle 1; as well as concentration (average) (Cavg), area under the curve from time 0 to the end of the dosing interval (Day 21) after repeated dosing (AUC0-τ), t1/2, clearance at steady state (CLss), volume of distribution during terminal phase (Vz), and accumulation ratio (Rac) (AUC0-τ/AUC0-21d) for longer-term analyses.

Tumor tissue samples will be collected in pre- and post-treatment for additional exploratory biomarkers. Tumor samples of Pre-treatment (i.e., Screening) could be obtained for c-Met status analysis by IHC through either subject's archived paraffin tissues or fresh (preferred) biopsies, and tumor tissue biopsies of post-treatment at C2D8 , pre- and post-treatments are optional. In addition, blood samples will also be collected in pre- and post-treatment and serum will be prepared for circulatory biomarker (soluble c-Met) analysis by ELISA at screening and C2D8; these blood samples are required in the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at both the Screening and baseline visits;
* Life expectancy ≥12 weeks
* Diagnosed (histologically or cytologically) with solid tumors and documented as advanced or metastatic disease for which there is no known effective anti-tumor treatment (refractory to or relapsed from standard therapies);
* Subjects must have measurable lesion(s) per RECIST v1.1 guideline at the Screening visit.
* Adequate laboratory parameters during the Screening Period as evidenced by:

  * Absolute neutrophil count (ANC)≥1.5×109/L (1,500/mm3)；
  * Platelets ≥100×109/L (100,000/mm3)；
  * Hemoglobin (Hgb) ≥9.0 g/dL (90 g/L)；
  * Albumin levels ≥2.8 g/dL；
  * Total bilirubin ≤1.5×ULN (≤3×ULN for subjects with liver metastases)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

    * 2.5×ULN; for subjects with liver metastases, ALT and AST ≤5×ULN；
  * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min based on Cockcroft-Gault equation；
* Subjects must have a washout period ≥4 weeks since the last dose of cytotoxic chemotherapy，non-cytotoxic chemotherapy(including any previous TKI treatment), any investigational therapy, any prior immuno-oncology or monoclonal antibody products administered and ≥6 weeks since the last dose of chemotherapy of mitomycin C or nitrosoureas prior to the first dose of SHR-A1403;
* Pregnancy and Contraception:

  * Female subjects agree not to be pregnant or lactating from beginning of the study screening until 6 months after receiving the last treatment;
  * Male and female subjects and their sexual partners are willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy from beginning of the study screening until 6 months after receiving the last treatment of study drug;
  * A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year, when used consistently and correctly);
  * Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of treatment and not be breast feeding. Female subjects of non-childbearing potential must be surgically sterile (i.e., bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing) OR naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing, with a follicle stimulating hormone (FSH) level at Screening of ≥40 mIU/mL;
* Willing and able to comply with clinic visits and study-related procedures;
* voluntarily participating in this clinical trial, understanding the study procedures and providing signed informed consent.

Exclusion Criteria:

* Known history of Grade 3 or Grade 4 hypersensitivity to any components (antibody-drug conjugate [ADC], total antibody, unconjugated toxin) of the SHR-A1403 product, or sensitivity to humanized monoclonal antibody products);
* Any radiation or surgery within 4 weeks prior to the first dose of SHR-A1403, except for minor palliative intent(this is to be discussed with sponsor);
* Unresolved toxicities from previous anticancer therapy,defined as toxicities not yet resolved to NCI CTCAE (current version) grade ≤1 at baseline (other than alopecia and other tolerable AEs upon discussion with sponsor) . Subjects with chronic grade 2 toxicities may be eligible at the discretion of the investigator and discussion with sponsor;
* Central nervous system tumors or active central nervous system (CNS) metastasis by imaging diagnosis;
* Cardiac disease (New York Heart Association [NYHA] classes II-IV) including myocardial infarction,unstable angina, congestive heart failure, or cardiac arrhythmia requiring treatment within a minimum 6 months before enrollment;
* Active HBV and HCV infection (HBV virus copy number>50 IU/mL, HCV virus RNA positive);
* History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV) or other acquired or congenital immune- deficient disease, or history of any organ transplantation;
* Any other medical(such as severe hypertension, diabetes, thyroid disease, etc.) or psychiatric or social condition deemed by the investigator to be likely serious hazards to a subject's rights, safety, welfare, or interfere with ability to sign informed consent, cooperate and participate in the study, interpret the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
The assessment of Treatment-related Adverse Events of SHR-A1403 in subjects with advanced solid tumors | up to 24 months
  Assessment of the incidence and severity of treatment-related Advanse events will be collected and analysed in all subjects who received at least 1 dose of SHR-A1403 with the current version of the NCI CTCAE
DLT | up to 24 months
  A DLT is considered at AE related to study drug unless there is a clear, well-documented, alternative explanation for the toxicity. Severity of AEs are graded according to the current version of the NCI CTCAE for the study, the occurence of the following drug related AEs during the first cycle(1 to 21days from the first infusion) will be considered a DLT by the investigator and SMC.
MTD | up to 24 months
  MTD is the highest dose whose toxicity probability was lower or close to the preset target level of toxicity probability (30% in this study) during the DLT observation in the dose escalation of SHR-A1403.

SECONDARY OUTCOMES:
Time to peak (Tmax) of serum concentration | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Time to peak (Tmax) of serum concentration
Maximum serum concentration (Cmax) | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Maximum serum concentration (Cmax)
Half-life (T1/2) | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Half-life (T1/2)
Clearance/ bioavailability (CL/F) | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Clearance/ bioavailability (CL/F)
Apparent volume of distribution/bioavailability (Vd/F) | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Apparent volume of distribution/bioavailability (Vd/F)
Area under curve (AUC) | Up to 24 months
  Pharmacokinetics profile of SHR-A1403:Area under curve (AUC)
Accumulation index (Rac) | up to 24 months
  Pharmacokinetics profile of SHR-A1403:Accumulation index (Rac)
The assessment of anti-drug antibody | up to 24 months
  The serum of patients who are administered with intravenous infusion every three weeks (q3w) for a treatment cycle are collected at difinitive time points， Anti-SHR-A1403 antibody will be detected and measured.
Preliminary efficacy assessments of SHR-A1403 | up to 24 months
  Subjects will be assessed every other cycle using RECIST v1.1.
C-Met expression levels in blood | up to 24 months
  The exploratory biomarker, C-Met,from blood samples obtained pre- and post-treatment will be measured.
C-Met expression levels in tumor tissue | up to 24 months
  The exploratory biomarker, C-Met, from tumor tissue samples obtained pre- and post-treatment will be measured.
The recommended Phase 2 dose (RP2D) of SHR-A1403 in subjects with advanced solid tumors | up to 24 months
  When the dose escalation is accomplished, RP2D will be reported by the assessment of safety with CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, China